CLINICAL TRIAL: NCT03686501
Title: An Open-Label Study To Evaluate D1 Receptor Occupancy (RO) Following a Single Dose of PF-06412562, Using Positron Emission Tomography (PET) With Ligand [18F]MNI-968 in Healthy Male Subjects
Brief Title: D1 Receptor Occupancy (RO) Following a Single Dose of PF-06412562
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F] MNI-968
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Healthy Male Volunteers
Keywords: HV

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06412562 (Experimental): To assess the D1 receptor occupancy (D1 RO) in striatum after a single oral administration of PF-06412562.
  Interventions: Drug: PF-06412562

INTERVENTIONS:
Drug: PF-06412562 — Healthy Volunteers recruited for the study will undergo a single dose of PF-06412562 and will undergo two [18F]MNI-968 injections
  Other Names: [18F]MNI-968 (PF-06730110)

SUMMARY:
To assess the D1 receptor occupancy (D1 RO) in striatum after a single oral administration of PF-06412562.

DETAILED DESCRIPTION:
Primary Objectives:

* To assess the D1 receptor occupancy (D1 RO) in striatum after a single oral administration of PF-06412562
* To assess the relationship of D1 RO in the striatum versus plasma exposure of PF-06412562 after a single oral administration.

Secondary Objective:

• To evaluate the plasma exposure of PF-06412562for the duration of PET scan following a single oral administration of PF-06412562.

Safety Objectives:

• To evaluate the safety and tolerability of PF-06412562 of single oral doses of PF-06412562.

ELIGIBILITY:
Inclusion Criteria:

Subject eligibility should be reviewed and documented by an appropriately qualified member of the investigator's study team before subjects are included in the study.

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study prior to the initiation of any study assessments.

   Healthy male subjects between the ages of 20 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests, in the opinion of the investigator).
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Male subjects must not donate sperm for the study duration.
4. Subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory test and other study procedures.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Evidence or history of clinically significant hepatic, renal, cardiovascular, endocrine, hematologic, gastrointestinal, pulmonary, neurologic, oncologic, psychiatric, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). This also includes subjects with previous history of epilepsy or seizures, clinically significant abnormal electroencephalogram (EEG), febrile convulsion, head injury with significant sequelae, psychiatric illness, attempted suicide or suicidal ideation.
2. Any condition possibly affecting drug absorption (eg, gastrectomy)
3. A positive urine drug screen (confirmed by repeat) Protocol 4006 Version 1.0; 20 April 2018 Confidential and Proprietary
4. History of regular alcohol consumption exceeding 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
5. Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the dose of study medication.
6. Screening supine blood pressure ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of rest. If blood pressure (BP) is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
7. 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
8. Males of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
9. Use of prescription drugs within 7 days or 5 half-lives (whichever is longer) prior to the dose of study medication. As an exception, acetaminophen/paracetamol may be used "as needed" (prn) and only at doses of ≤1 g/day.
10. Blood donation or loss (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
11. History of sensitivity to heparin or heparin-induced thrombocytopenia.
12. Unwilling or unable to comply with the Life Style Guidelines described in this protocol.
13. Any severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
14. A lifetime history of seizure disorder of any etiology, inclusive of childhood seizures.
15. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer or Invicro employees directly involved in the conduct of the study.
16. Use of drugs or consumption of foods/food products which inhibit CYP3A4 (including, but not limited to, atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, amprenavir, aprepitant, diltiazem, erythromycin, fluconazole, fosamprenavir, verapamil, cimetidine, grapefruit, grapefruit juice) within 7 days prior to the first dose of study medication.

    Protocol 4006 Version 1.0; 20 April 2018 Confidential and Proprietary
17. Evidence of orthostatic symptoms (eg, dizziness upon standing) or systolic blood pressure (BP) drop ≥20 mm Hg or diastolic BP drop ≥10 mm Hg from supine to standing assessment at screening. Abnormal values on Day 2 are left to the judgment of the investigator. Resting pulse rate < 45 or >100 bpm.
18. Any subject who is likely to be hospitalized (for any reason) during the study.
19. Subjects with pacemakers, aneurysm clips, artificial heart valves, ear implants, cerebrospinal fluid (CSF) shunts, metal fragments or foreign objects in the eyes, skin, or body, claustrophobia or any other condition that would contraindicate a brain MRI scan.
20. Inability to lie still within the environment of the MRI and PET scanners for the required period to acquire images.
21. Subjects with any anatomical abnormality in the head that would either preclude or tend to confound the analysis of study data, including any clinically significant abnormal findings from MRI of the head at screening.
22. Prior participation in other research protocols or clinical care within the past year in addition to the radiation exposure expected in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, equivalent with the acceptable annual limits established by the US Federal Guidelines.
23. Current, past or anticipated exposure to radiation for the past 5 years (for oncology-related radiation, refer to exclusion criteria #. This includes radiation therapy).
24. Subjects with a history of poor compliance history of refusing to comply with administered medications or inpatient/ research unit rules, or a history of demanding discharge from inpatient treatment against medical advice.
25. Subjects with screening laboratory test results that deviate from the upper or lower limits of the reference range, except for not clinically significant values, as determined by the investigator. Aspartate aminotransferase (AST) or Alanine transaminase (ALT) must be ≤2 X the upper limit of reference range, and total bilirubin must be within 1.5 X the upper limit of reference range at screening.
26. Subjects with a positive test for hepatitis B (HBsAg), hepatitis C antibody (HCV), Human Immunodeficiency Virus (HIV)1/HIV2 antibody/antigen.
27. Subjects who have answered "yes" to "Suicidal Ideation" Item 4 or Item 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Evaluate D1 Receptor Occupancy (RO) Following a Single Dose of PF-06412562, Using Positron Emission Tomography (PET) with Ligand [18F]MNI-968 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Invicro, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://www.invicro.com